CLINICAL TRIAL: NCT03969225
Title: Vascular Access Outcome Measure for Function: a vaLidation Study In haemoDialysis (VALID)
Brief Title: Vascular Access Outcome Measure for Function: a vaLidation Study In haemoDialysis
Acronym: VALID
Status: Completed | Type: Observational
Sponsor: The University of Queensland (Other)
Collaborators: Australasian Kidney Trials Network (Network)
Responsible Party: Sponsor
Other Study IDs: AKTN 19.01
Record Dates: First submitted 2019-05-10; First posted 2019-05-31 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2022-08

CONDITIONS: Vascular Access Complication; Hemodialysis Access Failure (Disorder)
Keywords: Haemodialysis vascular access; Core outcome; Vascular access function; Validation; Haemodialysis; Hemodialysis; Vascular access intervention; Vascular access procedure; Standardised outcomes in nephrology (SONG)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A functioning vascular access provides a lifeline for patients requiring haemodialysis but vascular access dysfunction remains one of the leading causes of excessive morbidity, mortality and healthcare costs in this group. Despite increasing numbers of vascular access trials, successful interventions to improve vascular access function have been sparse and compromised by highly variable, often selectively reported outcome measures of limited relevance to patients and health professionals. Through engagement of all relevant stakeholders including patients and caregivers, vascular access function, defined by the need for interventions to enable and maintain the use of a vascular access for haemodialysis, has been identified as one of the most critically important outcome measures for trials in haemodialysis. This prospective, multi-centre, multinational validation study aims to assess the accuracy and feasibility of measuring vascular access function part of routine clinical practice and across different clinical settings to ensure successful global implementation of this core outcome measure in future trials in haemodialysis.

DETAILED DESCRIPTION:
Haemodialysis is the most common treatment for patients with end-stage kidney disease worldwide and can only be provided via a functional vascular access. Patients, caregivers and health professionals consider vascular access function one of the most critically important outcomes in haemodialysis but trial-based evidence to improve vascular access function is limited by the inconsistent and selective reporting of this outcome. Reporting of a standardised outcome measure for vascular access function across all trials in haemodialysis will enhance the consistency and relevance of trial evidence to guide patient-centred care. Based on international contribution of all relevant stakeholders including patients, the need of interventions to enable and maintain the use of a vascular access for haemodialysis was considered a simple, pragmatic, and meaningful measure of vascular access function. To ensure global implementation across all trial in haemodialysis, it needs to be feasible to accurately collect this outcome measure as part of routine clinical practice without requiring additional resources or expertise in vascular access.

VALID is a prospective, multi-centre, multinational validation study to assess the accuracy and feasibility of measuring vascular access function, defined by the need for interventions to enable and maintain the use of a vascular access for haemodialysis by clinical staff as part of their routing clinical practice and across different clinical settings.

The primary objective of the VALID study is to determine whether vascular access function can be measured accurately by clinical staff as part of routine clinical practice compared to the reference standard of a research team with expertise in vascular access during a 6-month follow-up period.

An estimated 612 participants will be recruited from approximately 10 dialysis units of difference size, type (home-, in-centre and satellite), governance (private versus public), and location (rural versus urban) across Australia, Canada, China, France, United Kingdom, Netherlands, Malaysia and the United States of America (USA).

Implementation of a validated outcome measure for vascular access function across clinical trials will improve the reliability, comparability and relevance of future research in haemodialysis to inform patient-centred care.

ELIGIBILITY:
Inclusion Criteria:

* Patients new to or established on chronic haemodialysis (i.e. incident and prevalent patients on chronic haemodialysis)
* Patients 18 years or more of age
* Able to provide informed consent (if consent is required).

Exclusion Criteria:

* Anticipated to require haemodialysis for less than 90 days
* Treating team considers patient unsuitable to be enrolled
* Patient or authorised representative not willing to consent (if consent is required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving chronic haemodialysis in the participating unit and who are able and willing to provide informed consent, will be invited to take part in the trial. Patients who are expected to require haemodialysis for less than 3 months due to anticipated recovery of renal function will be excluded. The eligibility criteria are deliberately kept broad to reflect routine clinical practice (i.e. not excluding non-English speaking patients) and avoid selection bias within participating units. Paediatric patients are excluded because vascular access outcomes were not considered a core outcome domain for research in paediatric patients with chronic kidney disease as established by the SONG-Kids initiative involving children, adolescence, their family members, and health professionals.
Sampling Method: Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Reporting of vascular access function, defined by the need for any intervention(s) required to enable and maintain the use of a vascular access for haemodialysis. Vascular access interventions to be collected are outlined in the description below. | 6 months
  Arteriovenous fistula (AVF)/Arteriovenous graft (AVG)
  * Open surgical or endovascular creation/placement of AVF/AVG
  * Open surgical revision or endovascular intervention of AVG/AVF
  * Thrombolysis or thrombectomy of AVG/AVF
  * Ligation or resection of arteriovenous access
  * Repair of aneurysm/pseudoaneurysm
  * Competing/collateral vein ligation
  * Fistulogram (Angiogram) +/- angioplasty +/- stenting (including inflow artery, body of AVF/AVG, venous outflow, central vein)
  * Competing/collateral vein embolisation
  * Superficialisation/transposition
  * Management of Dialysis Associated Steal Syndrome (DASS)/Access Induced Ischaemia. Procedures include:
    * Distal Revascularisation, Interval Ligation (DRIL)
    * Proximalisation of the Arterial Inflow (PAI)
    * Revision Using Distal Inflow (RUDI)
    * Banding
  Central venous catheter (CVC)
  * CVC insertion
  * CVC exchange
  * Fibrin sheath removal/disruption
  * CVC removal

SECONDARY OUTCOMES:
Rate of vascular access interventions to enable and maintain the use of a vascular access for haemodialysis (number/patient-year). | 6 months
  Interventions collected as listed in the Primary Outcome description
Time to first vascular access intervention to enable and maintain the use of a vascular access for haemodialysis (days). | 6 months
  Interventions collected as listed in the Primary Outcome description
Type of vascular access interventions. | 6 months
  Interventions collected as listed in the Primary Outcome description

OTHER OUTCOMES:
Time required for measuring vascular access function (minutes) | 6 months
  Feasibility outcome measures
Completeness of data collection (percentage) | 6 months
  Feasibility outcome measures
Likert score of feasibility questionnaire with data collectors (scale of 1 to 5, 1=strongly disagree, 5=strongly agree) | 6 months
  Feasibility outcome measures
Qualitative analysis of semi structured interview with data collector | 6 months
  Feasibility outcome measures
Recruitment rate (number of participants/year) | 6 months
  Feasibility outcome measures
Eligibility ratio (number of patients eligible/number of patients screened) | 6 months
  Feasibility outcome measures
Enrolment ratio (number of patients enrolled/number of patients screened) | 6 months
  Feasibility outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Viecelli, MD, FRAC, Principal Investigator — Princess Alexandra Hospital and Australasian Kidney Trials Network
Locations (10):
- Australia (4):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Mackay Hospital, Mackay, Queensland
  - Mater Hospital, Brisbane
  - Hervey Bay Hospital, Hervey Bay
- University Health Network, Toronto, Canada
- Centre Hospitalier Régional Universitaire de Tours, Tours, France
- Hospital Sultanah Aminah Johor Bahru, Johor Bahru, Malaysia
- Maastricht University Medical Centre, Maastricht, Netherlands
- Ospedale Regionale di Lugano, Lugano, Switzerland
- Sheffield Teaching Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures and appendices) will be available for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: This process will be in effect for a period of 2 to 5 years following publication of the main study results. Proposals may be submitted up to 5 years following article publication. After 5 years, the data will be available in the Sponsor's data warehouse but without investigator support other than deposited metadata.
Access Criteria: An independent review board will assess proposals based on the following criteria: sound science, benefit-risk balancing and research team expertise.

REFERENCES:
- [Derived] Viecelli AK, Teixeira-Pinto A, Valks A, Baer R, Cherian R, Cippa PE, Craig JC, DeSilva R, Jaure A, Johnson DW, Kiriwandeniya C, Kopperschmidt P, Liu WJ, Lee T, Lok C, Madhan K, Mallard AR, Oliver V, Polkinghorne KR, Quinn RR, Reidlinger D, Roberts M, Sautenet B, Hooi LS, Smith R, Snoeijs M, Tordoir J, Vachharajani TJ, Vanholder R, Vergara LA, Wilkie M, Yang B, Yuo TH, Zou L, Hawley CM; VALID Investigator Team. Study protocol for Vascular Access outcome measure for function: a vaLidation study In hemoDialysis (VALID) : A multi-center, multinational validation study to assess the accuracy and feasibility of measuring vascular access function in clinical practice. BMC Nephrol. 2022 Nov 19;23(1):372. doi: 10.1186/s12882-022-02987-1. PMID 36402958
- See also: Enhancing the Quality and Transparency of health research (EQUATOR network). STARD 2015: An updated List of Essential Items for Reporting Diagnostic Accuracy Studies. — http://www.equator-network.org/reporting-guidelines/stard/
- See also: Standardised Outcomes in Nephrology (SONG) initiative. SONG-Haemodialysis Vascular Access Expert Working Group — http://songinitiative.org/projects/song-hd/song-hd-vascular-access/
- See also: Standardised Outcomes in Nephrology (SONG) Initiative. SONG Handbook (Version 1, 1st June 2017) for establishing and implementing core outcomes in chronic kidney disease. — http://songinitiative.org/reports-and-publications/